CLINICAL TRIAL: NCT00727506
Title: Phase I/II Trial of BIBW 2992 (Afatinib) in Treating Patients With Recurrent Glioblastoma Multiforme
Brief Title: BIBW 2992 (Afatinib) With or Without Daily Temozolomide in the Treatment of Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.36
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Afatinib; Temozolomide

ARMS (3):
- BIBW 2992 (Experimental): BIBW 2992 once daily
  Interventions: Drug: BIBW 2992
- TMZ (Active Comparator): TMZ 21/28 days
  Interventions: Drug: TMZ
- BIBW 2992 plus TMZ (Experimental): BIBW 2992 once daily plus TMZ 21/28 days
  Interventions: Drug: BIBW 2992 plus TMZ

INTERVENTIONS:
Drug: BIBW 2992 — BIBW 2992 once daily
  Arms: BIBW 2992
Drug: TMZ — TMZ 21/28
  Arms: TMZ
Drug: BIBW 2992 plus TMZ — BIBW 2992 once daily plus TMZ 21/28 days
  Arms: BIBW 2992 plus TMZ

SUMMARY:
Phase I Part: To determine the maximum tolerated dose (MTD) and pharmacokinetics of BIBW 2992 administered in combination with TMZ in patients with recurrent malignant gliomas (WHO Grade III and IV).

Phase II Part: To estimate the efficacy and safety of BIBW 2992 monotherapy and BIBW 2992 / TMZ combination therapy compared to TMZ monotherapy (three treatment arms) in patients with recurrent GBM. To evaluate molecular determinants of response to BIBW 2992.

ELIGIBILITY:
Inclusion criteria:

Phase I Part:

1. Histologically-confirmed WHO Grade III or IV malignant glioma that is recurrent after prior chemoradiotherapy. Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to WHO Grade III or IV malignant glioma.
2. Age at least 18 years at entry
3. KPS at least 60%
4. Patients must have recovered from previous surgery and chemotherapy.
5. Written informed consent that is consistent with local law and ICH-GCP guidelines.

Phase II Part:

1. Histologically-confirmed WHO Grade IV malignant glioma at first episode of recurrence after prior combined chemoradiotherapy. Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to WHO Grade IV malignant glioma and if prior treatment included temozolomide chemotherapy and radiotherapy.
2. Bi-dimensionally measurable disease with a minimum measurement of 1 cm (10 mm) in one diameter on Gd MRI performed within 14 days prior to first treatment (Day 1).
3. Age at least 18 years at entry
4. KPS at least 70%
5. Patients must have recovered from previous surgery and chemotherapy.
6. Written informed consent that is consistent with local law and ICH-GCP guidelines.
7. Patients receiving corticosteroids have to receive a stable or decreasing dose for at least 14 days before start of study treatment.

Exclusion criteria:

Phase I and Phase II Parts:

1. Less than 12 weeks between radiotherapy and start of study treatment, unless new enhancing lesion outside of radiation field or radiologically progressive on two consecutive MRI scans at least four weeks apart or biopsy-proven recurrence.
2. Less than two weeks from surgical resection (one week from prior stereotactic biopsy) or major surgical procedure.
3. Less than two weeks after previous chemotherapy (6 weeks from nitrosureas).
4. Treatment with other investigational drugs; participation in another clinical study within the past 2 weeks before start of therapy or concomitantly with this study.
5. Progressive disease or toxicity =CTCAEv3 Grade 3 to protracted temozolomide dosing (defined as temozolomide administered more than 5 days/28 day cycle).
6. Active infectious disease requiring intravenous therapy.
7. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
8. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea.
9. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
10. Patient is <3 years free of another primary malignancy except: if the other primary malignancy is either not currently clinically significant or does not require active intervention (such as a basal cell skin cancer or a cervical carcinoma in situ). Existence of any other malignant disease is not allowed.
11. Cardiac left ventricular function with resting ejection fraction <50%.
12. Absolute neutrophil count (ANC) less than 1500/mm3.
13. Platelet count less than 100,000/mm3.
14. Bilirubin greater than 1.5 x upper limit of institutional norm.
15. Aspartate amino transferase (AST) greater than 3 x upper limit of institutional norm.
16. Serum creatinine greater than 1.5 x upper limit of institutional norm.
17. Patients who are sexually active and unwilling to use a medically acceptable method of contraception.
18. Pregnancy or breast-feeding.
19. Patients unable to comply with the protocol.
20. Known pre-existing interstitial lung disease (ILD).

Phase I part only:

1. Less than four weeks from prior treatment with bevacizumab.

Phase II Part only:

1. Prior EGFR-directed therapy.
2. Prior bevacizumab therapy.
3. Patients presenting with second or higher number of episodes of recurrence.
4. Requirement of treatment with any of the prohibited concomitant medications listed in Section 4.2.2 (Restrictions regarding concomitant treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2008-07-14 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- United States (17):
  - 1200.36.0016 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1200.36.0012 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1200.36.0005 Boehringer Ingelheim Investigational Site, Duarte, California
  - 1200.36.0014 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1200.36.0019 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1200.36.0023 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1200.36.0008 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1200.36.0002 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1200.36.0003 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1200.36.0009 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.36.0001 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 1200.36.0007 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1200.36.0020 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1200.36.0017 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1200.36.0010 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1200.36.0011 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 1200.36.0022 Boehringer Ingelheim Investigational Site, Seattle, Washington
- Canada (11):
  - 1200.36.1005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1200.36.1010 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1200.36.1009 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1200.36.1011 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1200.36.1008 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1200.36.1001 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 1200.36.1003 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1200.36.1004 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1200.36.1007 Boehringer Ingelheim Investigational Site, Fleurimont, Quebec
  - 1200.36.1002 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1200.36.1006 Boehringer Ingelheim Investigational Site, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consists of 2 parts (phase I and phase II) with separate participants.
Groups:
- Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2: Patients receiving Afatinib 20mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part
- Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2: Patients receiving Afatinib 40mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part
- Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2: Patients receiving Afatinib 50mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part
- Phase II - Temozolomide 75mg/m^2: Patients receiving Temozolomide monotherapy 75 mg/m^2 for 21 days followed by 7 days off - Phase II part
- Phase II - Afatinib 40mg: Patients receiving Afatinib monotherapy 40mg once daily (q.d.) - Phase II part
- Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2: Patients receiving Afatinib 40mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase II part
Period: Overall Study
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2 | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Started | 6 (Entered) | 8 (Entered) | 18 (Entered) | 39 (Randomized) | 41 (Randomized) | 39 (Randomized)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 18 | 39 | 41 | 39
Not completed — Adverse Event | 0 | 0 | 4 | 4 | 1 | 8
Not completed — Dose Limiting Toxicity (DLT) | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Progressive disease | 4 | 7 | 9 | 28 | 38 | 28
Not completed — Refused to continue medication | 0 | 1 | 2 | 3 | 1 | 2
Not completed — Other reason not described above | 0 | 0 | 1 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: For Phase I part, all patients who were treated with at least one dose of the study medication. For Phase II part, all patients who were randomized and have taken at least one dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2 | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2 | Total
Number analyzed (Participants) | 6 | 8 | 18 | 39 | 41 | 39 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.4) | 51.6 (14.2) | 51.0 (9.4) | 56.9 (10.62) | 56.6 (9.44) | 55.4 (11.02) | 56.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 8 | 14 | 14 | 18 | 58
  Male | 4 | 6 | 10 | 25 | 27 | 21 | 93
Race/Ethnicity, Customized [Number; unit: Number of participants]
  Asian | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Black/African American | 0 | 0 | 2 | 2 | 0 | 2 | 6
  Hawaiian/Pacific Isle | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 6 | 7 | 16 | 37 | 40 | 35 | 141
Karnofsky performance score [Number; unit: Number of participants] — The scale range is from 100 (Normal no complaints) to 0 (dead). This score was used in Phase II randomization stratification and in some efficacy analyses.
  Number of participants
    70 | 1 | 1 | 1 | 9 | 9 | 12 | 33
    80 | 1 | 1 | 2 | 13 | 12 | 9 | 38
    90 | 2 | 4 | 11 | 12 | 17 | 15 | 61
    100 | 2 | 2 | 4 | 5 | 3 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With DLT- Phase I
Description: Number of Participants With Dose Limiting Toxicities (DLT) - Phase I Part
Time Frame: From randomization till data cut-off (10 Jun 2009), with a mean treatment duration of 51 days
Measure: Number; unit: participants
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2
Number analyzed (Participants) | 6 | 8 | 18
participants | 2 | 0 | 4

2. Primary Outcome: Progression-free Survival (PFS-6) at Six Months - Phase II
Description: PFS-6 is defined as probability of patients surviving to six months after randomization without progression. Disease progression was evaluated by an independent review committee and by the investigators, independently. The evaluation by the independent review committee was used for the primary outcome measure. The measurement "Number" the estimated PFS-6 value from the Kaplan-Meier curve of PFS.
Time Frame: At six months after randomization
Population: Randomised Set (RS). The randomised set includes all patients who were randomised to receive treatment in the Phase II part of the trial.
Measure: Number (95% Confidence Interval); unit: probablity of survival
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
probablity of survival | 0.230 [0.09 to 0.37] | 0.030 [0.00 to 0.09] | 0.103 [0.00 to 0.21]
Statistical Analysis 1: Comparison: Phase II - Temozolomide 75mg/m^2 vs Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2; Test type: Superiority or Other; p = 0.148, z-test — P-value is from an approximate normal test for the 6 month time point
Statistical Analysis 2: Comparison: Phase II - Temozolomide 75mg/m^2 vs Phase II - Afatinib 40mg; Test type: Superiority or Other; p = 0.008, z-test — P-value is an approximate normal test for the six month time point

3. Secondary Outcome: Objective Tumor Response in Phase I
Description: Objective Tumor Response is defined as complete response (CR) and partial response (PR) according to the MacDonald criteria assessed by central independent review.
Time Frame: From treatment start until the date of first documented progression or data cutoff at May 12, 2011, whichever came first, with a mean treatment duration of 69.7 days.
Population: Patients treated in Phase I part
Measure: Number; unit: participants
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2
Number analyzed (Participants) | 6 | 8 | 18
participants | 0 | 1 | 0

4. Secondary Outcome: Objective Tumor Response in Phase II
Description: Objective Tumor Response is defined as complete response (CR) and partial response (PR) according to the MacDonald criteria assessed by central independent review. Only data collected until cut-off date July 15, 2016 were considered.
Time Frame: From randomization to until the date of first documented progression or data cutoff on July 15, 2016, whichever came first, with a mean treatment duration of 110.0 days
Population: RS
Measure: Number; unit: participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
participants | 4 [2.9 to 24.2] | 1 [0.1 to 12.9] | 3 [1.6 to 20.9]
Statistical Analysis 1: Comparison: Phase II - Temozolomide 75mg/m^2 vs Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Phase II - Temozolomide 75mg/m^2 vs Phase II - Afatinib 40mg; Test type: Superiority or Other; p = 0.1954, Fisher Exact

5. Secondary Outcome: Progression-free Survival (PFS)- Phase II Part
Description: Progression-free survival was defined as the duration between randomization and the date of the first of the two following events: progression or death.
Time Frame: from date of randomization until the date of first documented progression or death by any cause, whichever came first, assessed up to 9 Months.
Population: Randomized set
Measure: Median (Full Range); unit: Months
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Months | 1.87 [1.15 to 3.68] | 0.99 [0.95 to 1.84] | 1.53 [0.99 to 1.87]
Statistical Analysis 1: Comparison: Phase II - Temozolomide 75mg/m^2 vs Phase II - Afatinib 40mg; Hazard ratio was calculated from Cox proportional hazard model stratified by age class (<=50 vs. >50 years old) and baseline Karnofsky Performance Scale (KPS) score (70, 80 vs. 90, 100). P-value was two-sided from log-rank test stratified by the same variables; Test type: Superiority or Other; p = 0.0320, Log Rank; Cox Proportional Hazard = 1.780, 95% CI 2-sided [1.088 to 2.912]
Statistical Analysis 2: Comparison: Phase II - Temozolomide 75mg/m^2 vs Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2; Hazard ratio was calculated from Cox proportional hazard model stratified by age class (<=50 vs. >50 years old) and baseline KPS score (70, 80 vs. 90, 100). P-value was two-sided from log-rank test stratified by the same variables; Test type: Superiority or Other; p = 0.2044, Log Rank; Cox Proportional Hazard = 1.392, 95% CI 2-sided [0.841 to 2.301]

6. Secondary Outcome: AUCτ,ss for Afatinib
Description: Area under the plasma concentration-time curve of afatinib after multiple administration (AUCτ,ss) of 50 mg afatinib in presence and absence of 75 mg/m² temozolomide (TMZ).
Time Frame: Before (-0.05 h) the drug administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8 h and 24 h after drug administration on Day 15 (in presence of temozolomide) and Day 28 (in absence of temozolomide) of treatment Cycle 1
Population: PKS Set and the patients who had enough PK samples for calculation of AUC. Pharmacokinetic set (PKS) : All patients who provided at least one blood sample were included in the Pharmacokinetic (PK) analysis.
Measure: Geometric Mean (Standard Deviation); unit: ng·h/mL
Groups:
- Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of TMZ): Patients receiving Afatinib 50mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part (in presence of temozolomide).
- Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of TMZ): Patients receiving Afatinib 50mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part (in absence of temozolomide).
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of TMZ) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of TMZ)
Number analyzed (Participants) | 15 | 5
ng·h/mL | 1070 (63.7) | 918 (65.3)

7. Secondary Outcome: Cmax,ss for Afatinib
Description: maximum measured plasma concentration of afatinib after multiple administration of 50 mg afatinib in presence and absence of 75 mg/m² temozolomide.
Time Frame: Before (-0.05 h) the drug administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8 h and 24h after drug administration on Day 15 (in presence of temozolomide) and Day 28 (in absence of temozolomide) of treatment Cycle 1
Population: PKS set
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of TMZ) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of TMZ)
Number analyzed (Participants) | 15 | 6
ng/mL | 63.2 (62.1) | 50.5 (58.0)

8. Secondary Outcome: Tmax,ss for Afatinib
Description: time from dosing to the maximum plasma concentration of afatinib after multiple administration of 50 mg afatinib in presence and absence of 75 mg/m² temozolomide
Time Frame: as for outcome 7
Population: PKS set
Measure: Median (Full Range); unit: hour
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of TMZ) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of TMZ)
Number analyzed (Participants) | 15 | 6
hour | 4.00 (58.0) [1.50 to 8.00] | 3.50 (62.1) [1.00 to 7.92]

9. Secondary Outcome: AUC (0-8) for Temozolomide
Description: Area under the plasma concentration-time curve over the time interval from zero to 08h (AUC (0-8)) of temozolomide in presence and absence of afatinib.
Time Frame: Before (-0.05 h) the first drug administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8 h after drug administration on Day 1 (in absence of afatinib) and Day 15 (in presence of afatinib) of treatment Cycle 1
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Groups:
- Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of Afatinib): Patients receiving Afatinib 50mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part (in presence of Afatinib).
- Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of Afatinib): Patients receiving Afatinib 50mg once daily (q.d.) plus Temozolomide 75 mg/m^2 for 21 days followed by 7 days off - Phase I part (in absence of Afatinib).
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of Afatinib) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of Afatinib)
Number analyzed (Participants) | 14 | 17
ng·h/mL | 8380 (24.1) | 8160 (27.8)

10. Secondary Outcome: Cmax for Temozolomide
Description: maximum measured plasma concentration following the first dose of uniform intervals τ (Cmax) of temozolomide in presence and absence of afatinib.
Time Frame: as for outcome 9
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of Afatinib) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of Afatinib)
Number analyzed (Participants) | 15 | 17
ng/mL | 2520 (33.3) | 2690 (39.7)

11. Secondary Outcome: Tmax for Temozolomide
Description: time from dosing to the maximum plasma concentration following the first dose of uniform intervals τ (tmax) of temozolomide in presence and absence of afatinib.
Time Frame: as for outcome 9
Population: PKS set
Measure: Median (Full Range); unit: h
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of Afatinib) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of Afatinib)
Number analyzed (Participants) | 15 | 17
h | 1.22 [1.00 to 3.25] | 1.00 [0.500 to 2.00]

12. Secondary Outcome: t1/2 for Temozolomide
Description: terminal half-life (t1/2) of temozolomide in presence and absence of afatinib
Time Frame: as for outcome 9
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Presence of Afatinib) | Phase I - Afatinib 50mg+TMZ 75mg/m^2 (in Absence of Afatinib)
Number analyzed (Participants) | 14 | 17
hours | 2.17 (34.3) | 2.08 (58.4)

13. Secondary Outcome: Phase II - Trough Plasma Concentration of Afatinib
Description: Trough plasma concentration of afatinib after multiple administration of 40 mg afatinib administered as monotherapy or in combination with 75 mg/m² temozolomide
Time Frame: Before (-0.05 h) the drug administration of afatinib on Day 15 of Cycle 2 & 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 41 | 39
ng/mL
  predose at Day 15 of Cycle 2 (n=17; 15) | 19.8 (69.5) [0.1 to 12.9] | 29.7 (72.1) [1.6 to 20.9]
  predose at Day 15 of Cycle 3 (n=10; 10) | 19.6 (70.8) | 20.2 (79.1)

14. Secondary Outcome: Number of Participants With EGFRvIII Assessed by IHC Test.
Description: Number of participants with the epidermal growth factor receptor variant III (EGFRvIII) assessed by IHC test for the evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for EGFRvIII by immunohistochemistry (IHC) test.
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  Sample tested: Negative | 6 | 8 | 5
  Sample tested: + | 5 | 3 | 4
  Sample tested: +/++ | 0 | 3 | 2
  Sample tested: ++ | 1 | 4 | 4
  Sample tested: ++/+++ | 1 | 3 | 3
  Sample tested: +++ | 3 | 5 | 10
  No Sample for test | 23 | 15 | 11

15. Secondary Outcome: Number of Participants With MGMT Marker Assessed by IHC Test.
Description: Number of participants with MGMT marker assessed by IHC test for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for O6-methylguanine-DNA methyltransferase (MGMT) by immunohistochemistry (IHC) test.
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  MGMT+ | 9 | 8 | 12
  MGMT- | 7 | 15 | 15
  No Sample for test | 23 | 18 | 12

16. Secondary Outcome: Number of Participants With EGFR Marker Assessed by IHC Test.
Description: Number of participants with EGFR marker assessed by IHC test for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for Epidermal Growth Factor Receptor (EGFR) by immunohistochemistry (IHC) test
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  EGFR wt+ | 14 | 23 | 24
  EGFR wt- | 2 | 0 | 4
  No Sample for test | 23 | 18 | 11

17. Secondary Outcome: Number of Participants With PTEN Marker Assessed by IHC Test.
Description: Number of participants with PTEN marker assessed by IHC test for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for Phosphatase and Tensin Homologue - a tumor suppressor gene/protein (PTEN) by immunohistochemistry (IHC) test.
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  PTEN intact | 5 | 4 | 7
  PTEN loss | 11 | 19 | 21
  No Sample for test | 23 | 18 | 11

18. Secondary Outcome: Number of Participants With PAKT Marker Assessed by IHC Test.
Description: Number of participants with PAKT marker assessed by IHC test for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for Serinethreonine kinase (PAKT) by immunohistochemistry (IHC) test.
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  PAKT+ | 5 | 11 | 11
  PAKT- | 11 | 13 | 16
  No Sample for test | 23 | 17 | 12

19. Secondary Outcome: Number of Participants With EGFR Assessed by FISH
Description: Number of participants with EGFR assessed by FISH for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for EGFR by fluorescent in situ hybridization (FISH).
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  EGFR abnormal (Amplification) | 5 | 14 | 11
  EGFR normal (Intact) | 1 | 0 | 1
  EGFR abnormal (Gain) | 10 | 9 | 16
  No Sample for test | 23 | 18 | 11

20. Secondary Outcome: Number of Participants With PTEN Assessed by FISH
Description: Number of participants with PTEN assessed by FISH for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for PTEN by fluorescent in situ hybridization (FISH).
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  PTEN abnormal (Loss) | 11 | 20 | 25
  PTEN normal (Gain) | 1 | 2 | 1
  PTEN normal (Intact) | 4 | 1 | 2
  No Sample for test | 23 | 18 | 11

21. Secondary Outcome: Number of Participants With Chromosomes (CEP7) Assessed by FISH
Description: Number of participants with Chromosomes (CEP7) assessed by FISH for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for Chromosomes (CEP7) by fluorescent in situ hybridization (FISH).
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  CEP7 abnormal (Gain) | 15 | 24 | 27
  CEP7 normal (Intact) | 1 | 0 | 1
  No Sample for test | 23 | 17 | 11

22. Secondary Outcome: Number of Participants With Chromosomes (CEP10) Assessed by FISH
Description: Number of participants with Chromosomes (CEP10) assessed by FISH for evaluation of molecular determinants of response to afatinib. Archival tumor samples from enrolled patients were collected and analyzed for Chromosomes (CEP10) by fluorescent in situ hybridization (FISH).
Time Frame: Baseline (during screening)
Population: Randomized set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  CEP10 abnormal (Loss) | 10 | 19 | 24
  CEP10 normal (Gain) | 2 | 3 | 1
  CEP10 normal (Intact) | 4 | 1 | 2
  No Sample for test | 23 | 18 | 11

23. Secondary Outcome: Number of Participants With Investigator Defined Drug-Related AEs, AEs Leading to Discontinuation of Trial Drug, All Serious Adverse Events (AE) and Other Significant AEs - Phase I
Description: Safety was assessed based on number of participants with investigator defined drug-related AEs, AEs leading to discontinuation of trial drug, All Serious Adverse events (AE) and other significant AEs (according to International Conference on Harmonisation (ICH) E3).
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 491 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2
Number analyzed (Participants) | 6 | 8 | 18
Participants
  drug-related AEs | 4 | 8 | 17
  AEs leading to discontinuation of trial drug | 2 | 1 | 10
  Serious AE's | 2 | 1 | 10
  other significant AEs | 1 | 0 | 5

24. Secondary Outcome: Number of Participants With Adverse Events (AEs) Based on Intensity and Incidence of AE's - Phase I
Description: Safety of afatinib as indicated by number of participants with adverse events based on intensity and incidence of AE's, especially skin reactions (rash, acne), gastrointestinal (GI) (Vomiting, nausea, diarrhea) and neurological
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 491 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2
Number analyzed (Participants) | 6 | 8 | 18
Participants
  Rash | 0 | 0 | 1
  Vomiting | 0 | 0 | 2
  Nausea | 0 | 1 | 0
  Diarrhoea | 0 | 1 | 2
  acne | 0 | 0 | 0
  Haemorrhage intracranial | 1 | 0 | 0
  Convulsion | 0 | 1 | 1
  Syncope | 0 | 1 | 0
  Hemiparesis | 0 | 0 | 2
  Aphasia | 0 | 0 | 1
  Brain oedema | 0 | 0 | 1
  Cerebrovascular accident | 0 | 0 | 1
  Headache | 0 | 0 | 1
  Paralysis | 0 | 0 | 1
  Peroneal nerve palsy | 0 | 0 | 1
  Vasogenic cerebral oedema | 0 | 0 | 1

25. Secondary Outcome: Number of Participants With Adverse Events, Graded According CTCAE - Phase I
Description: Safety of Afatinib assesed based on Number of participants with adverse events, graded according to United States National Cancer Institute Common terminology Criteria for Adverse Events (US NCI CTCAE) Version 3.0. The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 491 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2
Number analyzed (Participants) | 6 | 8 | 18
Participants
  Grade 1 | 1 | 2 | 0
  Grade 2 | 3 | 4 | 7
  Grade 3 | 0 | 1 | 7
  Grade 4 | 2 | 1 | 3
  Grade 5 | 0 | 0 | 1

26. Secondary Outcome: Causes of Death - Phase I
Description: Cause of the death reported during on treatment was due to disease progression.
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 491 days.
Population: Treated set
Measure: Number; unit: deaths
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2
Number analyzed (Participants) | 6 | 8 | 18
deaths | 0 | 0 | 1

27. Secondary Outcome: Number of Participants With Investigator Defined Drug-Related AEs, AE Leading to Dose Reduction, AEs Leading to Discontinuation of Trial Drug and All SAE- Phase II
Description: Safety was assessed based on number of participants with investigator defined drug-related AEs, AE leading to dose reduction, Adverse events (AEs) leading to discontinuation of trial drug and All Serious Adverse events (SAE).
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 518 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  drug-related AEs | 22 | 35 | 36
  AE leading to dose reduction | 2 | 4 | 7
  AEs leading to discontinuation of trial drug | 9 | 8 | 14
  Serious AE's | 6 | 10 | 13

28. Secondary Outcome: Number of Participants With Adverse Events (AEs) Based on Intensity and Incidence of AE's - Phase II
Description: as for outcome 24
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 518 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  Rash | 3 | 19 | 22
  Acne | 0 | 0 | 4
  Vomiting | 8 | 4 | 10
  Nausea | 7 | 6 | 13
  Diarrhoea | 4 | 29 | 32
  Neurological decompensation | 0 | 2 | 0
  Cerebral haemorrhage | 0 | 0 | 1
  Dysgeusia | 0 | 0 | 1
  Hemiparesis | 1 | 0 | 1
  Ataxia | 0 | 1 | 0
  Headache | 0 | 1 | 0
  Memory impairment | 0 | 1 | 0
  Speech disorder | 0 | 1 | 0

29. Secondary Outcome: Number of Participants With Adverse Events, Graded According CTCAE - Phase II
Description: Safety of Afatinib assessed based on the number of participants with adverse events, graded according to United States National Cancer Institute Common terminology Criteria for Adverse Events (US NCI CTCAE) Version 3.0. The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 518 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants
  Grade 1 | 3 | 5 | 2
  Grade 2 | 14 | 18 | 10
  Grade 3 | 13 | 15 | 19
  Grade 4 | 5 | 2 | 5
  Grade 5 | 2 | 1 | 2

30. Secondary Outcome: Causes of Death - Phase II
Description: Causes of death during on treatment.
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 518 days.
Population: Treated set
Measure: Number; unit: deaths
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
deaths
  Malignant Neoplasm Progression | 1 | 0 | 1
  Respiratory failure | 0 | 0 | 1
  Tumor progression | 1 | 1 | 0

31. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities for Decreased Cardiac Left Ventricular Function - Phase II
Description: Number of participants with Clinically Relevant Abnormalities for decreased Cardiac left ventricular function.
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 518 days.
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Number analyzed (Participants) | 39 | 41 | 39
Participants | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 491 days (Phase I) and 518 days (Phase II).
Arm/Group | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2 | Phase II - Temozolomide 75mg/m^2 | Phase II - Afatinib 40mg | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/8 | 10/18 | 6/39 | 10/41 | 13/39
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 18/18 | 36/39 | 40/41 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 (N=6) | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 (N=8) | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2 (N=18) | Phase II - Temozolomide 75mg/m^2 (N=39) | Phase II - Afatinib 40mg (N=41) | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2 (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Afatinib 20 mg Plus Temozolomide 75mg/m^2 (N=6) | Phase I - Afatinib 40 mg Plus Temozolomide 75mg/m^2 (N=8) | Phase I - Afatinib 50 mg Plus Temozolomide 75mg/m^2 (N=18) | Phase II - Temozolomide 75mg/m^2 (N=39) | Phase II - Afatinib 40mg (N=41) | Phase II - Afatinib 40mg Plus Temozolomide 75 mg/m^2 (N=39)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 5 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 3 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 4 | 7 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 13 | 4 | 29 | 31
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 8 | 6 | 13
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 7 | 8 | 4 | 8
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 4
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 4 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 3 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 3 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 0 | 7
Weight increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 3 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 5 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 7 | 2 | 1 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 4 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3 | 3 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 4
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 3 | 1
Aphasia (Nervous system disorders) | 1 | 1 | 0 | 6 | 2 | 4
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 4 | 3 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 5 | 2 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 4
Headache (Nervous system disorders) | 2 | 0 | 2 | 10 | 6 | 10
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 4 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 6 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 1 | 4 | 3
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 4 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 3 | 2 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 4 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 3 | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 2 | 3 | 3 | 3
Depression (Psychiatric disorders) | 0 | 1 | 2 | 1 | 2 | 5
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 4 | 2
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 4 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 4 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0 | 6 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3 | 9
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 5 | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 7 | 13 | 3 | 18 | 22
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 3 | 2 | 1 | 4
Chills (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Fatigue (General disorders) | 1 | 2 | 9 | 10 | 9 | 11
Gait disturbance (General disorders) | 0 | 0 | 1 | 4 | 3 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 4 | 4
Oedema peripheral (General disorders) | 0 | 0 | 1 | 4 | 3 | 4
Temperature intolerance (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2 | 9 | 3
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
White blood cells urine (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 2 | 1 | 3 | 0 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.